CLINICAL TRIAL: NCT05337124
Title: A Prospective Observational Registry of Patients Treated With LUPKYNIS® (Voclosporin) in the US
Acronym: ENLIGHT-LN
Status: Completed | Type: Observational
Sponsor: Aurinia Pharmaceuticals Inc. (Industry)
Collaborators: United BioSource, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: AUR-VCS-2021-03
Record Dates: First submitted 2022-03-22; First posted 2022-04-20 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — voclosporin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lupkynis Treatment Group
  Interventions: Drug: LUPKYNIS

INTERVENTIONS:
Drug: LUPKYNIS — LUPKYNIS treatment per the approved US Prescribing Information
  Other Names: voclosporin

SUMMARY:
This registry is an observational study designed to assess the utilization and effectiveness of LUPKYNIS in adult patients with lupus nephritis (LN) in the United States (US).

DETAILED DESCRIPTION:
This registry is an observational study designed to assess the utilization and effectiveness of LUPKYNIS in patients with lupus nephritis (LN) in the United States (US). This registry is intended to benefit and support interests of patients, clinicians, regulatory bodies, payers, and industry by obtaining longitudinal data on LUPKYNIS.

ELIGIBILITY:
Inclusion Criteria:

* Lupus nephritis (LN) confirmed by biopsy
* Initiating or have initiated treatment with commercial LUPKYNIS as per US approved Prescribing Information (PI)
* Written informed consent

Exclusion Criteria:

- Off-label use (Use of LUPKYNIS outside of the FDA-approved US Prescribing Information)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All lupus nephritis patients that meet the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
LUPKYNIS utilization patterns | 12 months (1 year) to 60 months (5 years)
  The proportion of patients that had their first Urine Protein Creatinine Ratio (UPCR) >0.5 mg within 6 months of initiating LUPKYNIS.
Effectiveness of LUPKYNIS | 12 months (1 year) to 60 months (5 years)
  The proportion of patients that achieve Urine Protein Creatinine Ratio (UPCR) <=0.5 mg after initiating LUPKYNIS by race, ethnicity, and previous LN treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Aurinia Study Director, Study Director — Aurinia Pharmaceuticals Inc.
Locations (1):
- Site 00-05, South Gate, California, United States

IPD SHARING:
Plan to Share IPD: No